CLINICAL TRIAL: NCT02180581
Title: Effect of Probiotics in Reducing Infections and Allergies in Young Children Starting Daycare
Acronym: ProbiComp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: The Danish Council for Strategic Research (Other); Chr Hansen A/S (Unknown); Technical University of Denmark (Other); University of Bergen (Other); Odense University Hospital (Other); Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-4-2014-032; H-4-2014-032 (Other Grant/Funding Number: The Danish Council for Strategic Research)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Days Absent From Daycare; Respiratory Tract Infections; Gastrointestinal Infections; Allergy
Keywords: Infections; Allergy; Immune function; Microbiota; Infant
MeSH Terms: conditions — Respiratory Tract Infections; Hypersensitivity; Infections | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (2 * 10^9 cfu/d) (Experimental): Daily intake of bifidobacterium animalis ssp. Lactis (BB12) and Lactobacillus Rhamnosus GG (LGG) in a dosage of 10^9 cfu/day of each strain. The probiotics are provided as powder in a sachet, and can be added to food or drink
  Interventions: Dietary Supplement: Probiotic (2 * 10^9 cfu/day)
- Placebo (Placebo Comparator): provided as powder in a sachet, and can be added to food or drink
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic (2 * 10^9 cfu/day) — Combination of two probiotics (2 * 10^9 cfu/day) or probiotics for 6 months
  Other Names: bifidobacterium animalis ssp. Lactis (BB12), 10^9 cfu/day; Lactobacillus Rhamnosus GG (LGG), 10^9 cfu/day
  Arms: Probiotic (2 * 10^9 cfu/d)
Dietary Supplement: Placebo — Placebo for 6 months
  Arms: Placebo

SUMMARY:
The aim of the intervention is to examine the effect of a combination of the two bacterial strains BB-12 and LGG, provided for 6 month, on the prevalence of infections and allergic manifestations in small children, and how a combination of BB-12 and LGG affects the immune system, gastrointestinal tract and the microbiota. Children are enrolled during 2 winter seasons.

ELIGIBILITY:
Inclusion Criteria:

* Expected to start daycare between the age of 8-14 month
* Intervention start 0 days to 12 weeks before starting daycare
* Expected to start daycare from september to february (both month included)
* Single born

Exclusion Criteria:

* Exclusion Criteria:
* Children born before 37th gestational week
* Children with a birth weight < 2500 g
* Children suffering from severe chronic illness
* Children receiving regular medication
* Children who have received antibiotics within a month before intervention start
* Children whose parents do not speak Danish

Ages: 8 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 290 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of days absent from daycare due to respiratory and gastrointestinal infections | up to 6 month
  Recorded weekly by the parents using web-based questionnaires

SECONDARY OUTCOMES:
Acute upper respiratory tract infections | Up to 6 month
  Number of days with acute upper respiratory tract infections (URTI); Number of children with at least 1 episode of URTI; Number of children with at least 3 episodes of URTI; Number of URTI episodes/child/year; Duration of URTI episodes (days);
  Additionally,symptoms of cold (defined as 2 days with runny/stuffy nose or cough)
  Recorded by the parents daily/weekly using web-based questionnaires.
Acute lower respiratory infections | Up to 6 month
  Number of children with at least 1 episode of a lower respiratory tract infection (LRTI).
  LRTI include bronchitis and pneumonia
  Recorded by the parents weekly using web-based questionnaires.
Gastrointestinal infections | Up to 6 month
  Number of children with at least 1 episode of diarrhea; Duration of episodes with diarrhea(days); Number of episodes/child/year with diarrhea; Number of days with vomiting.
  Recorded by the parents daily using web-based questionnaires
Fever | Up to 6 month
  Number of days with fever
  Recorded by the parents using web-based questionnaires
Antibiotic use | Up to 6 month
  Number of treatments with antibiotics during the intervention period
  Recorded weekly by the parents using web-based questionnaires
Allergies | Up to 6 month
  Number of children developing allergies during the intervention period (asthma, allergic rhinitis, atopic dermatitis, food allergies); Age for diagnosis of allergies; Use of medication due to allergies.
  Recorded by the parents using web-based questionnaires
Absence from day care due to illness other than infections | Up to 6 month
  Number of days the child is absent from day care due to illness, which is not due to infections.
  Recorded by the parents weekly using web-based questionnaires
Parental absence from work due to illness of the child | Up to 6 month
  Number of days a parent is absent from work due to illness of the child (infections and other illnesses, respectively)
  Recorded by the parents weekly using web-based questionnaires
Medical visits | Up to 6 month
  Number of visits to a doctor due to infections and other illnesses, respectively.
  Recorded by the parents using web-based questionnaires
Change from baseline in Thymus size | At baseline and after 6 mo (end of intervention)
  Change in thymic size during intervention period will be evaluated using ultrasound

OTHER OUTCOMES:
Change from baseline in biological markers for the immune system | At baseline and after 6 mo
  Analysis of biological material investigating the effect on the immune system by biological markers .
Change from baseline in biological markers for gastro-intestinal tract | At baseline and after 6 mo
  Analysis of biological material investigating the effect on the gastrointestinal tract.
Change from baseline in Biological markers of allergy | At baseline and after 6 mo
  analysis of biological samples investigating the effect on allergy by biological markers at baseline and at 6 mo

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Paediatric and International Nutrition, Department of Nutrition, Exercise and Sports, Faculty of Science, University of Copenhagen, Frederiksberg, Denmark

REFERENCES:
- [Derived] Schmidt RM, Pilmann Laursen R, Bruun S, Larnkjaer A, Molgaard C, Michaelsen KF, Host A. Probiotics in late infancy reduce the incidence of eczema: A randomized controlled trial. Pediatr Allergy Immunol. 2019 May;30(3):335-340. doi: 10.1111/pai.13018. Epub 2019 Feb 21. PMID 30790361
- [Derived] Laursen MF, Laursen RP, Larnkjaer A, Michaelsen KF, Bahl MI, Licht TR. Administration of two probiotic strains during early childhood does not affect the endogenous gut microbiota composition despite probiotic proliferation. BMC Microbiol. 2017 Aug 17;17(1):175. doi: 10.1186/s12866-017-1090-7. PMID 28818050